CLINICAL TRIAL: NCT02282917
Title: Exploratory Evaluation of AR-42 Histone Deacetylase Inhibitor in the Treatment of Vestibular Schwannoma and Meningioma
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Drug manufacturing logistics; lack of access to drug supply
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: Johns Hopkins University (Other); Stanford University (Other); Ohio State University (Other); Nationwide Children's Hospital (Other); Mayo Clinic (Other)
Responsible Party: Principal Investigator, D. Bradley Welling, MD, PhD, Chief Otolaryngology Massachusetts Eye and Ear, Massachusetts Eye and Ear Infirmary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-078H
Record Dates: First submitted 2014-10-31; First posted 2014-11-05 (Estimated); Results first posted 2022-05-11 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2021-12

CONDITIONS: Vestibular Schwannoma; Meningioma; Acoustic Neuroma; Neurofibromatosis Type 2
Keywords: NF2; Vestibular Schwannoma; Schwannoma; Meningioma
MeSH Terms: conditions — Neuroma, Acoustic; Meningioma; Neurofibromatosis 2; Neurilemmoma | interventions — HDAC-42

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AR-42 Administration (Experimental): AR-42 will be administered three times per week beginning 3 weeks prior to surgery.
  Interventions: Drug: AR-42

INTERVENTIONS:
Drug: AR-42 — AR-42 will be administered in a total of ten oral doses, +/- 1 dose, at 40 mg/dose, will be self-administered by study participants at approximately 8:00pm (+/- 1 hour) for 3 weeks pre-operatively, with the last dose being administered the night before surgery. The treating surgeon will perform the clinically indicated surgical procedure 3 weeks post-initial dose of medication as well as the specimen collection.
  Other Names: OSU-HDAC42

SUMMARY:
This will be a multi-center, proof of concept phase 0 study to assess the suppression of p-AKT in Vestibular Schwannoma (VS) and meningiomas by AR-42 in adult patients undergoing tumor resection. AR-42 is a small molecule which crosses the blood brain barrier (BBB) in rodents, but the investigators are not certain yet if it will penetrate human VS. Meningiomas are outside the BBB, but seem to be unusually resistant to all current medical treatments. The primary endpoint of the bioactivity of suppression of p-AKT by AR-42 was selected as drug activity seems more informative than bioavailability. Our preclinical data and others have shown dose dependent suppression of p-AKT by AR-42 in both VS and meningiomas.

DETAILED DESCRIPTION:
This is a multi-center, proof of concept phase 0 study to assess the suppression of p-AKT in VS and meningiomas by AR-42 in adult patients undergoing NF2-tumor resection. AR-42 will be administered three times per week beginning 3 weeks prior to surgery. A total of ten doses, +/- 1 dose at 40 mg/dose, will be self-administered orally by study participants at approximately the same time every day (+/- 1 hour, preferably in the evening) 3 times per week for 3 weeks pre-operatively, with the last dose taken the night before surgery. Patients will be evaluated within the context of their standard post-operative follow up which includes within 2 days of surgery and again at 2 weeks (+/- 10 days) after surgery. Samples will be shipped to the participating laboratories (OSU Comprehensive Cancer Center (CCC) Pharmacoanalytical Shared Resource (PhASR) and Nationwide Children's Research Institute) for assessment of intratumoral drug concentration and assessment of intratumoral disease markers. During surgery, four blood samples will also be obtained and sent to the cooperating laboratory (PhASR) for determination of drug concentration and molecular analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with vestibular schwannoma and/or meningioma diagnosed by MRI where surgical resection has been selected as treatment.
* Patients diagnosed with NF2 must meet Manchester Criteria.
* Age > 18 years of age
* Prior biologic therapy, chemotherapy, surgery or radiation is permitted.
* At the time of screening, the patient must have normal organ and marrow function.
* Eastern Cooperative Oncology Group/World Health Organization (ECOG/WHO) performance status of 0-1.
* Patients must be able to swallow capsules.
* Patients or their legal representatives must be able to read, understand and provide informed consent to participate in the trial.
* Tumor type will be confirmed by a neuropathologist.
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL prior to starting AR-42.
* The patient must be willing to comply with fertility requirements

Exclusion Criteria:

* Pregnant women are excluded from this study because the potential for teratogenic or abortifacient effects of AR-42 are not known. Because there is an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother with AR-42, breastfeeding should be discontinued if the mother is treated with AR-42.
* Pediatric patients are excluded from the phase 0 study as the effects of AR-42 are not known on children and there is no potential direct benefit to them.
* Patients with malabsorption or any other condition that in the opinion of the principal investigator could cause difficulty in absorption of drug.
* Patients requiring chronic corticosteroids (dose equivalent > 20mg prednisolone).
* Concurrent use of complementary or alternative medicines that in the opinion of the principal investigator would confound the interpretation of toxicities and/or antitumor activity of the study drug.
* Patients with a "currently active" second malignancy that, in the opinion of the principal investigator, will interfere with patient participation, increase patient risk, or confound data interpretation.
* Patients with a mean QTcB > 450 msec in males and > 470 msec in females.
* Patients with long QT syndrome.
* Patients who are being treated for an active infection.
* Patients receiving the following concomitant medications:

  * Any other anti-neoplastic chemotherapy or biologic therapy during the study
  * Concomitant radiotherapy
  * Concomitant HDAC inhibitors (e.g. valproic acid) as class-specific adverse reactions may be additive
  * Use of granulocyte colony-stimulating factors including G-CSF, pegylated G-CSF or GM-CSF should follow ASCO guidelines for patients receiving anti-cancer therapy.
  * Drugs associated with QT/QTc prolongation (see Appendix A)
* Patients who are receiving concurrent anti-neoplastic therapy.
* Any other medical condition, including mental illness or substance abuse, deemed by the principal investigator to likely interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.
* Patients with significant cardiovascular disease, including a myocardial infarction or unstable angina within 6 months or unstable cardiac arrhythmias are not eligible for the study.
* Known HIV infection, as their immunosuppressive conditions may complicate potential pancytopenias seen with HDAC inhibitors and complicate evaluation of drug effect.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2021-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad Welling, MD, PhD, Principal Investigator — Massachusetts Eye and Ear
Locations (4):
- United States (4):
  - Stanford University, Stanford, California
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts Eye and Ear, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Welling DB, Collier KA, Burns SS, Oblinger JL, Shu E, Miles-Markley BA, Hofmeister CC, Makary MS, Slone HW, Blakeley JO, Mansouri SA, Neff BA, Jackler RK, Mortazavi A, Chang LS. Early phase clinical studies of AR-42, a histone deacetylase inhibitor, for neurofibromatosis type 2-associated vestibular schwannomas and meningiomas. Laryngoscope Investig Otolaryngol. 2021 Aug 20;6(5):1008-1019. doi: 10.1002/lio2.643. eCollection 2021 Oct. PMID 34667843
- [Derived] Cheng H, Xie Z, Jones WP, Wei XT, Liu Z, Wang D, Kulp SK, Wang J, Coss CC, Chen CS, Marcucci G, Garzon R, Covey JM, Phelps MA, Chan KK. Preclinical Pharmacokinetics Study of R- and S-Enantiomers of the Histone Deacetylase Inhibitor, AR-42 (NSC 731438), in Rodents. AAPS J. 2016 May;18(3):737-45. doi: 10.1208/s12248-016-9876-3. Epub 2016 Mar 4. PMID 26943915

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seven participants were identified and recruited by the study investigators and/or study coordinators within the Department of Otolaryngology at Massachusetts Eye and Ear, Boston, MA. Participants were identified by their clinical history with vestibular schwannomas, meningiomas, cutaneous schwannomas, and/or Neurofibromatosis Type 2. The first enrollment took place in December 2015, and the final enrollment took place in July 2017.
Pre-assignment Details: Following all participant enrollments (consent), baseline procedures to determine eligibility included: complete blood count with differential and platelets, comprehensive metabolic panel, coagulation panel (PT/PTT), chest x-ray, neurological exam, pregnancy testing, 12-lead ECG, audiogram, and MRI (CPT 70553). Participants were terminated from the study after their baseline visit if they did not meet all eligibility requirements.
Groups:
- AR-42 Administration: There was no randomization in this trial and all participants completed study procedures uniformly. AR-42 was administered three times per week beginning 3 weeks prior to surgery. AR-42 was administered in a total of ten oral doses, +/- 1 dose, at 40 mg/dose, which was self-administered by study participants at approximately 8:00pm (+/- 1 hour) for 3 weeks pre-operatively, with the last dose being administered the night before surgery. All participants were instructed to take the study medication at least 1 hour before, or 2 hours after, a meal. The principal investigator performed the clinically indicated surgical procedure 3 weeks post-initial dose of medication as well as the specimen collection.
Period: Overall Study
Arm/Group | AR-42 Administration
Started | 7
Completed | 5
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Screen Failure/Not Eligible | 1

BASELINE CHARACTERISTICS:
Population: Two participants were withdrawn from the study prior to the administration of the study drug: one was deemed ineligible, and one chose not to participate.
Groups:
- AR-42 Administration: AR-42 was administered three times per week beginning 3 weeks prior to surgery. AR-42 was administered in a total of ten oral doses, +/- 1 dose, at 40 mg/dose, and was self-administered by study participants at approximately 8:00pm (+/- 1 hour) for 3 weeks pre-operatively, with the last dose being administered the night before surgery. A study investigator performed the clinically indicated surgical procedure 3 weeks post-initial dose of medication as well as the specimen collection.
Arm/Group | AR-42 Administration
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 54.9 [30 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
Weight [Mean (Full Range); unit: kilograms (kg)] — Population: Two participants were withdrawn from the study prior to baseline weight measurement.
  kilograms (kg) | 98.22 [82.6 to 120.0]
Prior tumor biopsy or debulking [Count of Participants; unit: Participants]
  Yes | 0
  No | 5
Relevant diagnosis [Count of Participants; unit: Participants]
  Sporadic vestibular schwannoma | 4
  Sporadic meningioma | 1
ECOG Grade [Count of Participants; unit: Participants] — The ECOG Scale of Performance Status grades a patient's level of functioning in terms of their ability to care for themselves and other activities of daily living. Grading is done from 0 (zero) to 5 (five). An ECOG grade of 0 (zero) is defined as "fully active, able to carry on all pre-disease performance without restriction." An ECOG grade of 4 (four) is defined as "completely disabled; cannot carry on any selfcare; totally confined to bed or chair." An ECOG grade of 5 (five) is defined as death.
  Participants
    ECOG = 0 | 4
    ECOG not assessed at baseline | 1
Baseline plasma concentration of AR-42 [Mean (Full Range); unit: nanomolar (nM)] — Population: Plasma concentrations of AR-42 at baseline (before tumor resection) are reported individually for each of the 5 participants.
  nanomolar (nM)
    number analyzed (Participants) | 1
    (all) | 150.18 [3.5 to 362.3]

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Phospho-AKT (p-AKT) to AKT After 3 Weeks of Oral AR-42
Description: The phospho-AKT/AKT ratio was used to estimate the activity of AKT, a kinase, at the core of resected tumors. Quantitation of the normalized p-AKT/AKT ratio is depicted as a percentage relative to the untreated VS2 set as 100%. For example, a value under 100% indicates a lower level of AKT activity relative to untreated VS2 tumors. Phosphorylated AKT, or phospho-AKT, is the activated form of AKT. These measurements were derived from the core of the resected tumors.
Time Frame: 3 weeks
Measure: Mean (Full Range); unit: percent (%)
Arm/Group | AR-42 Administration
Number analyzed (Participants) | 5
percent (%) | 53.6 [19 to 105]

2. Primary Outcome: Peripheral Phospho-AKT (p-AKT) to AKT Ratio After 3 Weeks of Oral AR-42
Description: The phospho-AKT/AKT ratio was used to estimate the activity of AKT, a kinase, at the core of resected tumors. Quantitation of the normalized p-AKT/AKT ratio is depicted as a percentage relative to the untreated VS2 set as 100%. For example, a value under 100% indicates a lower level of AKT activity relative to untreated patients. Phosphorylated AKT, or phospho-AKT, is the activated form of AKT. These measurements were derived from the periphery of the resected tumors.
Time Frame: 3 weeks
Measure: Mean (Full Range); unit: percent (%)
Arm/Group | AR-42 Administration
Number analyzed (Participants) | 5
percent (%) | 61.2 [9 to 102]

3. Secondary Outcome: AR-42 Plasma Concentration
Description: Steady-state plasma concentrations of AR-42 at the time of tumor resection are provided.
Time Frame: 1 week
Measure: Mean (Full Range); unit: nanomolar (nM)
Arm/Group | AR-42 Administration
Number analyzed (Participants) | 5
nanomolar (nM) | 107.58 [3.4 to 303.7]

4. Secondary Outcome: AR-42 Tumor Concentration (Capsule)
Description: Concentrations of AR-42 at the tumor capsule are provided.
Time Frame: 1 week
Measure: Mean (Full Range); unit: nanomolar (nM)
Arm/Group | AR-42 Administration
Number analyzed (Participants) | 5
nanomolar (nM) | 325.1 [16.2 to 5296.6]

5. Secondary Outcome: AR-42 Tumor Concentration (Center)
Description: Intra-tumor concentrations of AR-42 at the tumor center are reported.
Time Frame: 1 week
Measure: Mean (Full Range); unit: nanomolar (nM)
Arm/Group | AR-42 Administration
Number analyzed (Participants) | 5
nanomolar (nM) | 645.18 [7.1 to 1766.2]

6. Secondary Outcome: AR-42 Tumor Concentration (Capsule/Plasma)
Description: Capsule/plasma intra-tumor AR-42 concentrations are provided as a ratio.
Time Frame: 1 week
Measure: Mean (Full Range); unit: ratio
Arm/Group | AR-42 Administration
Number analyzed (Participants) | 5
ratio | 13.078 [1.72 to 53.4]

7. Secondary Outcome: AR-42 Tumor Concentration (Center/Plasma)
Description: Center/plasma intra-tumoral AR-42 concentrations are provided as a ratio.
Time Frame: 1 week
Measure: Mean (Full Range); unit: ratio
Arm/Group | AR-42 Administration
Number analyzed (Participants) | 5
ratio | 5.748 [1.59 to 17.8]

8. Other Pre Specified Outcome: Number of Doses of AR-42 Received
Description: We report the average total number of doses of AR-42 taken per participant during this study.
Time Frame: 3 weeks
Measure: Median (Full Range); unit: total doses
Arm/Group | AR-42 Administration
Number analyzed (Participants) | 5
total doses | 9 [8 to 11]

ADVERSE EVENTS:
Time Frame: Participants were observed for adverse events over 5 weeks, beginning 3 weeks prior to surgery and ending 2 weeks after surgery. This interval included perioperative adverse events and surgical complications associated with AR-42.
Description: Adverse events were graded according to Common Terminology Criteria for Adverse Events (CTCAE) and were also recorded according to severity, expectedness, and relatedness to the investigational treatment. Participants were encouraged throughout the study to spontaneously report all adverse events promptly to their physician-investigator.
Arm/Group | AR-42 Administration
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AR-42 Administration (N=5)
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Fatigue (General disorders) | 3
Nausea (General disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 1
Confusion (Psychiatric disorders) | 4
Lymphopenia (Blood and lymphatic system disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Taste change (Nervous system disorders) | 1
Headache (General disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 2
Facial weakness (Nervous system disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 2
Non-cardiac chest pain (General disorders) | 2
CSF leak (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 1
Scleral disorder (Eye disorders) | 1

LIMITATIONS AND CAVEATS:
The supplier of AR-42 was unable to continue to supply drugs after 2017. We elected to present the data on five of the originally planned 20 patients. Accrual was also limited by patient willingness to accept potential additional peri-operative risk without a reasonable likelihood of benefit from only 3 weeks of therapy with AR-42. Other limitations include possible selection bias, lack of control subjects, and the inability to perform meaningful statistical analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT02282917/Prot_SAP_000.pdf